# Advantages of Single-port Laparoscopy in the Treatment of Benign Ovarian Tumors in Children and Adolescents: A Multicenter Retrospective Study October 1, 2023

## Advantages of Single-port Laparoscopy in the Treatment of Benign Ovarian Tumors in Children and Adolescents: A Multicenter Retrospective Study

- 1. Starting and ending date of the project study: January 2019 to January 2023
- 2. Introduction of research content:

A multi-center analysis was performed on children and adolescents with benign ovarian tumors in 6 hospitals in Fujian province, and the removal of benign ovarian tumors by porous laparoscopy or ovarian cysts by single-pore laparoscopy was performed to analyze the incidence and clinical characteristics of gynecologic tumors in children and adolescents. The operation time, intraoperative blood loss, intraoperative tumor rupture rate, anal exhaust time, hospital stay, aesthetic score (CS) and visual analogue score (VAS) were compared between the two groups.

#### 3. Research objectives:

To compare the efficacy of single-aperture laparoscopy and porous laparoscopy in benign ovarian tumors in Chinese children and adolescents, and to explore the most suitable minimally invasive surgical treatment for this special population, so as to guide clinical practice.

#### 4. Research design and methods:

1) Data collection: Data of multicenter patients meeting the criteria were collected, and their general clinical data, including age, diagnosis, pathology, and ovarian tumor size (mean tumor diameter; In the case of bilateral ovaries, the diameter of the larger

side was recorded), location of ovarian tumor, operation time, intraoperative blood loss, and intraoperative tumor rupture rate. In addition, postoperative complications, anal exhaust time, length of hospital stay, cosmetic score, VAS score, and 5-point Likert satisfaction Scale were collected.

2) Statistical analysis: Clinical characteristics, surgery-related indicators, postoperative pain and aesthetic satisfaction of patients in the two groups were compared by statistical methods.

#### 5. Inclusion and exclusion criteria:

Inclusion criteria: ① patients ≤18 years old; ② Postoperative pathological diagnosis confirmed benign ovarian tumor; ③ Multi-hole laparoscopic or single-hole laparoscopic surgery; ④ Medical records and pathological data were complete and available.

Exclusion criteria: ① Patients with malignant pathological diagnosis; ② Patients undergoing open surgery; ③ Incomplete medical records or pathological data.

### 6. Protection measures for subjects:

The medical records used in this study were obtained from previous clinical diagnosis and treatment, and the postoperative satisfaction of patients was interviewed by telephone. The researchers would inform the information orally and obtain the consent of patients and their families before the study. By controlling the risk of disclosure of personal privacy through anonymization and other means, the subject will not accept any additional medical intervention/examination, will not increase the risk of routine

diagnosis and treatment, will not affect his access to normal medical services, and the risk to the subject is less than the minimum risk. Any public reporting of the results of this study will not identify the individual patients. We will make every effort to protect the privacy of our patients' personal medical information to the extent permitted by law.